CLINICAL TRIAL: NCT01311973
Title: Assessment of the Relationship Between Salivary Phosphorus and Level of Kidney Function
Brief Title: Salivary Phosphorus and Level of Kidney Function
Status: Completed | Type: Observational
Sponsor: Denver Nephrologists, P.C. (Other)
Collaborators: CM&D Pharma Limited (Industry)
Responsible Party: Geoffrey A. Block, MD, Principal Investigator, Denver Nephrologists, P.C.
Other Study IDs: CMD 003
Record Dates: First submitted 2011-03-03; First posted 2011-03-10 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease, phosphorus, salivary phosphorus
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, and saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Renal Function Group #1: Creatinine clearance > 90 mL/min
- Renal Function Group #2: Creatinine clearance 60-69 mL/min
- Renal Function Group #3: Creatinine clearance 50-59 mL/min
- Renal Function Group #4: Creatinine clearance 40-49 mL/min
- Renal Function Group #5: Creatinine clearance 30-39 mL/min
- Renal Function Group #6: Creatinine clearance 20-29 mL/min
- Renal Function Group #7: Creatinine clearance < 20 mL/min (not on dialysis)

SUMMARY:
The specific purpose of this study is to describe the relationship between salivary phosphorus and kidney function, specifically as it relates to serum phosphorus, FGF23, PTH, vitamin D status and urinary excretion of phosphorus.

DETAILED DESCRIPTION:
Previous studies have demonstrated that salivary phosphate levels are elevated in patients with chronic kidney disease and that there is a direct and linear correlation between serum phosphorus and salivary phosphorus. However, data regarding the relationship between salivary phosphate levels and stage of kidney disease (estimated glomerular filtration rate (eGFR) is lacking; as such, this study seeks to examine that relationship.

There is a normal circadian rhythm to serum phosphorus with a mid-afternoon peak at approximately 3 PM and a nadir at approximately 7-11 AM. Furthermore it has been demonstrated that a fasting serum phosphorus level at 8 AM is NOT indicative of 24 hour mean serum phosphorus. Thus the relationship between salivary phosphorous and serum phosphorus may vary over the course of the day.

This is a single-center study in which saliva, urine, and serum will be collected at two time points in a minimum of 105 subjects with various degrees of renal function (not on dialysis). Assignment to the renal group will be based upon the Visit 2 estimated glomerular filtration rate value. Enrollment in each group will continue at random until the target of 15 subjects per group is achieved. It is possible that an individual group may exceed the target enrollment number as their assignment will occur retrospectively.

All subjects will be required to have their morning assessment conducted between the hours of 7AM and 11AM. Clinical chemistry, serum phosphorus, intact parathyroid hormone(iPTH), plasma fibroblast growth factor 23 (FGF-23),serum 1,25 di-hydroxyvitamin D, serum 25-OH vitamin D, and a spot urine will be collected. A 24-hour urine sample will also be collected.

Passive and stimulated salivary collection will occur. The salivary collection must occur in a fasting state with nothing to eat or drink for at least 90 minutes prior to the collection.

Subjects will be permitted to leave the facility. They will be instructed to consume a lunch of their choice between the hours of 1100AM and 1200PM. They will be instructed to eat nothing after 1200PM. Subjects will return to the clinic for Visit 3 as directed by the study staff. Visit 3 will be conducted between 1PM and 4PM. Laboratory assessments, salivary collections, and spot urines will be collected at Visit 3. A dietary recall of intake at Visit 2 and 3 will also be completed.

ELIGIBILITY:
Inclusion Criteria:

* Men or women greater than 18 years of age.
* The subject has voluntarily signed and dated the most recent informed consent form approved by an Institutional Review Board (IRB).

Exclusion Criteria:

* Receiving hemodialysis.
* Receiving or has received an investigational product (or is currently using an investigational device) within 28 days prior to Visit 2.
* Evidence of active and clinically significant infection at Visit 2.
* Dental work within 48 hours prior to Visit 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal healthy population an individuals with chronic kidney disease not on dialysis
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Correlation between fasting salivary phosphorus and estimated glomerular filtration rate | single value between 7-11 am
  subjects with various levels of estimated glomerular filtration rate will have a single assessment in the fasted state of salivary phosphorus
Correlation between post meal salivary phosphorus and estimated glomerular filtration rate | single value after meal between 1-4 pm
  subjects with various levels of estimated glomerular filtration rate will have a single assessment in the fed state (meal between 11 am - 12 noon) of salivary phosphorus measured between 1-4 pm

SECONDARY OUTCOMES:
correlation of fasting salivary phosphorus with plasma fibroblast growth factor 23 levels(FGF-23) | single AM measurement between 7-11 am
  subjects will have plasma FGF23 measured in the fasting state between 7-11 am and correlation made with simultaneous assessment of salivary phosphorus
Correlation between fasting salivary phosphorus and serum 1,25 vitamin D levels. | single AM measurement between 7-11 am
  subjects will have serum 1,25 vitamin D measured in the fasting state between 7-11 am and correlation made with simultaneous assessment of salivary phosphorus
Correlation between fasting salivary phosphorus and serum intact parathyroid hormone (iPTH) levels. | single AM measurement between 7-11 am
  subjects will have serum intact parathyroid hormone measured in the fasting state between 7-11 am and correlation made with simultaneous assessment of salivary phosphorus

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrologists, PC
Locations (1):
- Denver Nephrologists, PC, Denver, Colorado, United States

REFERENCES:
- [Derived] Block GA, Persky MS, Shamblin BM, Baltazar MF, Singh B, Sharma A, Pergola P, Smits G, Comelli MC. Effect of salivary phosphate-binding chewing gum on serum phosphate in chronic kidney disease. Nephron Clin Pract. 2013;123(1-2):93-101. doi: 10.1159/000351850. Epub 2013 Jun 22. PMID 23797006